CLINICAL TRIAL: NCT06308224
Title: Comparison of Modified-Otago and Tai Chi Exercises on Balance and Motor Function in Patients With Stroke
Brief Title: Comparison of Modified-Otago and Tai Chi Exercises in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0290
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Modified-Otago Exercises; Tai-Chi Exercises; Stroke; Randomized Clinical Trial
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single-blinded as the assessor of the study would be kept blind of the treatment groups to which the patient would be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Modified-Otago Exercises) (Experimental): Participants will engage in Modified-Otago exercises for 30 minutes of moderate-intensity exercise at least three times weekly for 12 weeks.
  1. Walking for 15 minutes
  2. Strengthening exercises for 10 minutes
  3. Balance exercises 20 minutes
  Interventions: Other: Modified-Otago Exercises
- Group B (Tai Chi Exercises) (Experimental): Participants of the Tai Chi qigong group will participate in a 30-minute exercise class three times a week for 12 weeks.
  1. Warm-up exercises for 10 minutes
  2. Tai Chi Exercises for 30 minutes
  3. Cool-down exercises for 5 minutes
  Interventions: Other: Tai-Chi Exercises

INTERVENTIONS:
Other: Modified-Otago Exercises — Walking for 15 minutes before or after the strengthening and balance exercises of Modified-Otago.
  Strengthening exercises for 10 minutes: Knee extensor, Knee flexor, Hip adductor, Ankle plantar flexors (calf raises), and Ankle dorsiflexion (toe raises).
  Balance exercises 20 minutes: Knee bends, Backwards walking, Walking and turning around, Sideways walking, Tandem stance (heel-toe stand), Tandem walk (heel-toe walk), One leg stand, Heel walking, Toe walk, Heel toe walking backward, sit to stand and Stair walking.
  Other Names: Rehabilitation
  Arms: Group A (Modified-Otago Exercises)
Other: Tai-Chi Exercises — Warm-up exercises for 10 minutes.
  Tai Chi Qigong Exercises for 30 minutes: Commencing form and regulating breathing, Expanding your chest, Painting a rainbow, Circling arms to separate the clouds, Fixed step invert brachial, Row a boat in the middle of the lake, Shoulder the ball, Turning the body to look at the moon, Twisting waist and pushing palms, Horse step and cloud hands, Drag the sea and watch the sky, Undulating waves, Dove spreading wings, Extend arms and punch, Wild goose flying, Flywheel turning, Bounce ball while stepping, Pressing palms in calmness.
  Cool-down exercises for 5 minutes.
  Other Names: Rehabilitation
  Arms: Group B (Tai Chi Exercises)

SUMMARY:
The study aims to determine the comparative effects of Modified-Otago and Tai Chi Exercises on Balance and Motor Function in Patients with Stroke.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at the Physiotherapy and Chiropractor Centre, Lahore. Data will be collected within seven months after the approval of synopsis. A total of 64 patients will be recruited through convenience sampling technique after inclusion and exclusion criteria. After the baseline assessment, randomizations will be performed through the lottery method. Group A will receive Modified Otago exercises for 60 minutes, 3 times per week for 12 weeks, and Group B will receive Tai Chi Qigong exercises for 60 minutes, 3 times per week for 12 weeks. To assess the balance and motor function, the Berg Balance Scale (BBS) and Motor Assessment Scale will be used, respectively. The data will be analyzed by using the SPSS (Statistical Package for Social Sciences) 23 version.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed stroke patients with ischemic type.
2. Post-stroke ≥ 3 months.
3. Survivors of both hemorrhagic and ischemic stroke.
4. Subjects should have stable conditions after the stroke incidence.
5. Community-dwelling survivors of stroke who were aged ≥40 years.
6. Both genders can participate in the study.
7. Mini-Mental State Exam score equal to or greater than 24.
8. Modified Rankin Scale score of three or less.
9. Berg Balance Scale score is between 41 and 52.
10. Muscle strength grade should be of grade 4 and above.

Exclusion Criteria:

1. Subjects with diagnosed peripheral neuropathy.
2. The subject is unable to perform Tai Chi exercises.
3. No history of other neurological and musculoskeletal conditions.
4. Subjects with diagnosed vestibular disease.
5. Subjects have cardiac abnormalities.
6. Contracture, fracture, or pain in the musculoskeletal system.
7. Subjects who have undergone strength and balance training in the past 3 months.
8. Subject taking medications that increase the incidence of falls.
9. Subjects have been diagnosed with malignancy of any type.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 12 weeks
  The BBS, a 14-item scale, quantitatively evaluates balance and fall risk in older community-dwelling adults by directly observing their performance. Scores range from 0 to 4, with 0 indicating inability and 4 representing independent completion. The total score, out of 56, categorizes balance as impaired (0-20), acceptable (21-40), or good (41-56).
Timed Up and Go (TUG) | 12 weeks
  The Timed Up and Go (TUG) is a comprehensive physical performance test designed to evaluate mobility, balance, and locomotor abilities in elderly individuals dealing with balance issues. The test involves a sequence of motor tasks related to walking and turning. Without specific items, the individual is required to stand up from a chair (not leaned against a wall), walk 3 meters, turn around, return to the chair, and sit down at a comfortable pace.
Motor Assessment Scale (MAS) | 12 weeks
  The Motor Assessment Scale (MAS) serves as a performance-based evaluation tool designed to assess everyday motor function in stroke patients. It encompasses 8 items representing different areas of motor function. A single item assesses the general tonus to estimate muscle tone on the affected side. Ratings, scored on a 7-point scale (0-6), indicate optimal motor behavior, with a sum of item scores (excluding general tonus) providing an overall score out of 48 points.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No